CLINICAL TRIAL: NCT05034380
Title: Epigenetic Effects of a Single Bout of Exercise on Cardiovascular Risk Factors and the Metabolome in Lean and Overweight or Obese Subjects
Brief Title: Epigenetic Effects of a Single Bout of Exercise on Cardiovascular Risk Factors and the Metabolome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Purdue University (Other); Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Jessica Ellis, Assistant Professor, East Carolina University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AcuteExerciseNucleo
Record Dates: First submitted 2020-09-16; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Type 2 Diabetes; Cardiovascular Diseases; Acute Exercise
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All participants underwent the same exact study protocol on random days throughout the study period.
Who Masked: Outcomes Assessor
Masking Description: Investigators conducting molecular analysis were blinded to study samples/groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean (Active Comparator): males aged 18-30 years with BMI < 25
  Interventions: Behavioral: Acute exercise
- Overweight/Obese (Experimental): males aged 18-30 years with BMI >= 25
  Interventions: Behavioral: Acute exercise

INTERVENTIONS:
Behavioral: Acute exercise — All participants consumed a standardized, high carbohydrate meal (7 kcal/kg; 60% carbohydrate, 25% fat, 15% protein) and completed an exercise testing trial, expending a total of 650 kcal upon completion 4h later.

SUMMARY:
The purpose of this study is to determine the ability of acute exercise to regulate fat metabolism in muscle of overweight and obese people compared to lean people.

DETAILED DESCRIPTION:
After being informed about the study details and possible risks and benefits, 15 overweight/obese and 15 lean participants gave written informed consent and were then screened and enrolled in the study. All participants then gave a muscle sample and ate a calorically controlled breakfast. Participants completed ~1 hour of cycling exercise on a stationary bike and gave a second muscle sample 4 hours after eating breakfast.

ELIGIBILITY:
Inclusion Criteria:

* healthy males that completed a physical examination with a State Licensed M.D. or D.O. within the past 2 years and completed a physical activity readiness questionnaire (PARQ), the International Physical Activity Questionnaires (IPAQ) and and a medical history questionnaire prior to the study

Exclusion Criteria:

* any participants that had not had a physical examination by a State Licensed M.D. or D.O. within the past 2 years
* persons not considered "healthy" (with any previous medical diagnoses) or not medically cleared by a M.D. or D.O. to perform physical activity/exercise
* persons who are regularly physically active

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09-14 (Actual); Primary Completion 2015-10-06 (Actual); Study Completion 2016-03-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in skeletal muscle acylcarnitines | Baseline and immediately after acute cycling exercise
  Metabolomics of skeletal muscle acylcarnitines is used as a measure of mitochondrial function by assessing long, medium and short chain acylcarnitine levels.
Change from baseline in skeletal transcriptome | Baseline and immediately after acute cycling exercise
  RNA-seq is a method used to quantify changes in all known messenger RNA levels in the genome, giving an assessment of whole genome gene transcription changes.
Change from baseline in skeletal muscle whole genome nucleosome maps | Baseline and immediately after acute cycling exercise
  MNase-seq is a method used to determine the occupancy/location of nucleosomes throughout the entire genome, supporting evidence of alterations in epigenetic modifications occurring at specific genomic loci that affect nucleosome occupancy/location and possibly gene transcription or silencing.

SECONDARY OUTCOMES:
Glucose | Baseline and immediately after acute cycling exercise
  Commercially validated and available colorimetric used to determine plasma glucose levels.
Insulin | Baseline and immediately after acute cycling exercise
  Commercially validated and available ELISAs used to determine plasma insulin levels.
Triglycerides | Baseline and immediately after acute cycling exercise
  Commercially validated and available colorimetric kits used to determine plasma triglyceride levels.
Free fatty acids | Baseline and immediately after acute cycling exercise
  Commercially validated and available colorimetric kits used to determine plasma free fatty acid levels.
Cholesterol | Baseline and immediately after acute cycling exercise
  Commercially validated and available colorimetric kits used to determine total cholesterol, HDL, LDL and VLDL levels in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Henagan, PhD, Principal Investigator — Purdue University, Louisiana State University Medical School at Shreveport
Locations (1):
- Purdue University, West Lafayette, Indiana, United States